CLINICAL TRIAL: NCT04121052
Title: A Phase 1, 4-Period, Crossover, Open-label Study in Healthy Volunteers to Assess the Effect of Different Types of Food on a Single-dose of JNJ-64417184 Administered as Tablets
Brief Title: A Study in Healthy Volunteers to Assess the Effect of Different Types of Food on a Single-dose of JNJ-64417184 Administered as Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR108707; 2019-003469-17 (EudraCT Number); 64417184RSV1006 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-10-08; First posted 2019-10-09 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Treatment Sequence 1 (Experimental): Participants will receive JNJ-64417184 oral tablet in fed conditions (high-fat meal) in treatment period 1; followed by JNJ-64417184 oral tablet in fed conditions (low-fat meal) in treatment period 2; followed by JNJ-64417184 oral tablet in fed conditions (Ensure Original) in treatment period 3; followed by JNJ-64417184 oral tablet in fed conditions (standard meal) in treatment period 4, on Day 1 of each treatment period. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-64417184
- Treatment Sequence 2 (Experimental): Participants will receive JNJ-64417184 oral tablet in fed conditions (low-fat meal) in treatment period 1; followed by JNJ-64417184 oral tablet in fed conditions (standard meal) in treatment period 2; followed by JNJ-64417184 oral tablet in fed conditions (high-fat meal) in treatment period 3; followed by JNJ-64417184 oral tablet in fed conditions (Ensure Original) in treatment period 4, on Day 1 of each treatment period. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-64417184
- Treatment Sequence 3 (Experimental): Participants will receive JNJ-64417184 oral tablet in fed conditions (standard meal) in treatment period 1; followed by JNJ-64417184 oral tablet in fed conditions (Ensure Original) in treatment period 2; followed by JNJ-64417184 oral tablet in fed conditions (low-fat meal) in treatment period 3; followed by JNJ-64417184 oral tablet in fed conditions (high-fat meal) in treatment period 4, on Day 1 of each treatment period. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-64417184
- Treatment Sequence 4 (Experimental): Participants will receive JNJ-64417184 oral tablet in fed conditions (Ensure Original) in treatment period 1; followed by JNJ-64417184 oral tablet in fed conditions (high-fat meal) in treatment period 2; followed by JNJ-64417184 oral tablet in fed conditions (standard meal) in treatment period 3; followed by JNJ-64417184 oral tablet in fed conditions (low-fat meal) in treatment period 4, on Day 1 of each treatment period. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-64417184
- Treatment Sequence 5 (Experimental): Participants will receive JNJ-64417184 oral tablet in fed conditions (high-fat meal) in treatment period 1; followed by JNJ-64417184 oral tablet in fed conditions (low-fat meal) in treatment period 2; followed by JNJ-64417184 oral tablet under fasted condition in treatment period 3; followed by JNJ-64417184 oral tablet in fed conditions (standard meal) in treatment period 4, on Day 1 of each treatment period. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-64417184
- Treatment Sequence 6 (Experimental): Participants will receive JNJ-64417184 oral tablet in fed conditions (low-fat meal) in treatment period 1; followed by JNJ-64417184 oral tablet in fed conditions (standard meal) in treatment period 2; followed by JNJ-64417184 oral tablet in fed conditions (high-fat meal) in treatment period 3; followed by JNJ-64417184 oral tablet under fasted condition in treatment period 4, on Day 1 of each treatment period. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-64417184
- Treatment Sequence 7 (Experimental): Participants will receive JNJ-64417184 oral tablet in fed conditions (standard meal) in treatment period 1; followed by JNJ-64417184 oral tablet under fasted condition in treatment period 2; followed by JNJ-64417184 oral tablet in fed conditions (low-fat meal) in treatment period 3; followed by JNJ-64417184 oral tablet in fed conditions (high-fat meal) in treatment period 4, on Day 1 of each treatment period. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-64417184
- Treatment Sequence 8 (Experimental): Participants will receive JNJ-64417184 oral tablet under fasted condition in treatment period 1; followed by JNJ-64417184 oral tablet in fed conditions (high-fat meal) in treatment period 2; followed by JNJ-64417184 oral tablet in fed conditions (standard meal) in treatment period 3; followed by JNJ-64417184 oral tablet in fed conditions (low-fat meal) in treatment period 4, on Day 1 of each treatment period. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-64417184
- Treatment Sequence 9 (Experimental): Participants will receive JNJ-64417184 oral tablet in fed conditions (high-fat meal) in treatment period 1; followed by JNJ-64417184 oral tablet in fed conditions (low-fat meal) in treatment period 2; followed by JNJ-64417184 oral tablet under fasted condition in treatment period 3; followed by JNJ-64417184 oral tablet in fed conditions (Ensure Original) in treatment period 4, on Day 1 of each treatment period. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-64417184
- Treatment Sequence 10 (Experimental): Participants will receive JNJ-64417184 oral tablet in fed conditions (low-fat meal) in treatment period 1; followed by JNJ-64417184 oral tablet in fed conditions (Ensure Original) in treatment period 2; followed by JNJ-64417184 oral tablet in fed conditions (high-fat meal) in treatment period 3; followed by JNJ-64417184 oral tablet under fasted condition in treatment period 4, on Day 1 of each treatment period. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-64417184
- Treatment Sequence 11 (Experimental): Participants will receive JNJ-64417184 oral tablet in fed conditions (Ensure Original) in treatment period 1; followed by JNJ-64417184 oral tablet under fasted condition in treatment period 2; followed by JNJ-64417184 oral tablet in fed conditions (low-fat meal) in treatment period 3; followed by JNJ-64417184 oral tablet in fed conditions (high-fat meal) in treatment period 4, on Day 1 of each treatment period. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-64417184
- Treatment Sequence 12 (Experimental): Participants will receive JNJ-64417184 oral tablet under fasted condition in treatment period 1; followed by JNJ-64417184 oral tablet in fed conditions (high-fat meal) in treatment period 2; followed by JNJ-64417184 oral tablet in fed conditions (Ensure Original) in treatment period 3; followed by JNJ-64417184 oral tablet in fed conditions ( low-fat meal) in treatment period 4, on Day 1 of each treatment period. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-64417184
- Treatment Sequence 13 (Experimental): Participants will receive JNJ-64417184 oral tablet in fed conditions (high-fat meal) in treatment period 1; followed by JNJ-64417184 oral tablet in fed conditions (standard meal) in treatment period 2; followed by JNJ-64417184 oral tablet under fasted condition in treatment period 3; followed by JNJ-64417184 oral tablet in fed conditions (Ensure Original) in treatment period 4, on Day 1 of each treatment period. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-64417184
- Treatment Sequence 14 (Experimental): Participants will receive JNJ-64417184 oral tablet in fed conditions (standard meal) in treatment period 1; followed by JNJ-64417184 oral tablet in fed conditions (Ensure Original) in treatment period 2; followed by JNJ-64417184 oral tablet in fed conditions (high-fat meal) in treatment period 3; followed by JNJ-64417184 oral tablet under fasted condition in treatment period 4, on Day 1 of each treatment period. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-64417184
- Treatment Sequence 15 (Experimental): Participants will receive JNJ-64417184 oral tablet in fed conditions (Ensure Original) in treatment period 1; followed by JNJ-64417184 oral tablet under fasted condition in treatment period 2; followed by JNJ-64417184 oral tablet in fed conditions (standard meal) in treatment period 3; followed by JNJ-64417184 oral tablet in fed conditions (high-fat meal) in treatment period 4, on Day 1 of each treatment period. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-64417184
- Treatment Sequence 16 (Experimental): Participants will receive JNJ-64417184 oral tablet under fasted condition in treatment period 1; followed by JNJ-64417184 oral tablet in fed conditions (high-fat meal) in treatment period 2; followed by JNJ-64417184 oral tablet in fed conditions (Ensure Original) in treatment period 3; followed by JNJ-64417184 oral tablet in fed conditions (standard meal) in treatment period 4, on Day 1 of each treatment period. A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: JNJ-64417184

INTERVENTIONS:
Drug: JNJ-64417184 — Participants will receive single dose of JNJ-64417184 as oral tablet.

SUMMARY:
The purpose of this study is to evaluate the effect of 5 different food conditions on the single dose pharmacokinetics (PK) of the JNJ-64417184 tablet formulation administered orally, using the PK after a high-fat meal as a reference, in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Must have a body mass index (BMI); weight per height square between 18.0 and 30.0 kilogram per meter square (kg/m^2), (extremes included), and body weight not less than 50.0 kg at screening
* Healthy on the basis of physical examination, medical and surgical history, and vital signs performed at screening. If there are abnormalities, the participant may be included only if the investigator judges the abnormalities to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Must have a normal 12-lead electrocardiogram (ECG) (triplicate) at screening, including: normal sinus rhythm (heart rate between 45 and 100 beats per minute [bpm], extremes included); QT interval corrected for heart rate (QTc); QRS interval less than (<) 120 milliseconds (ms); PR interval less than or equals to <= 200 ms. If the results of the ECG are outside the normal ranges, the subject may be included only if the investigator judges the deviations from normal ECG to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the subject's source documents and initialed by the investigator
* Female participant must have a negative highly sensitive serum beta human chorionic gonadotropin (Beta-hCG) pregnancy test at screening and on Days -1 for each treatment period (except for postmenopausal female participants)
* Must not use nicotine-containing substances including tobacco products (example, cigarettes, e-cigarettes, cigars, chewing tobacco, gum, or patch) for at least 3 months prior to screening

Exclusion Criteria:

* Any evidence of heart block or bundle branch block at screening
* Current human immunodeficiency virus (HIV)-type 1 (HIV-1) or HIV-2 infection (confirmed by antibodies) at screening
* History of hepatitis A, B, or C infection, or current hepatitis A infection (confirmed by hepatitis A antibody immunoglobulin M [IgM]), or HBV infection (confirmed by hepatitis B surface antigen), or HCV infection (confirmed by HCV antibody) at screening
* A history of clinically significant drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy witnessed in previous studies with experimental drugs
* Has previously been dosed with JNJ-64417184

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Plasma Concentration of JNJ-64417184 under Fasted and Fed (Low-fat meal, Ensure Original, Standard meal, and High-Fat Meal as a Reference) Conditions | Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 72, 96, 120 hours postdose
  Plasma concentration of JNJ-64417184 under fasted and fed (low-fat meal, Ensure Original, standard meal, and high-fat meal as a reference) conditions will be determined.

SECONDARY OUTCOMES:
Plasma Concentration of JNJ-64417184 under Fasted and Fed (Low-fat meal, Ensure Original, Standard meal, Excluding High-fat Meal) Conditions | Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 72, 96, 120 hours postdose
  Plasma Concentration of JNJ-64417184 under Fasted and Fed (low-fat meal, Ensure Original, standard meal, and excluding high-fat meal) conditions will be determined.
Maximum Observed Analyte Concentration (Cmax) of JNJ-64417184 | Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 72, 96, 120 hours postdose
  Cmax is the maximum observed analyte concentration.
Area Under the Concentration-time Curve from Time Zero to the Last Measurable Concentration (AUC [0-last]) of JNJ-64417184 | Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 72, 96, 120 hours postdose
  AUC (0-last) is area under the plasma analyte concentration- time curve (AUC) from time 0 to time of the last quantifiable (non-below quantification limit [non-BQL]) concentration, calculated by linear-linear trapezoidal summation.
Area Under the Concentration-time Curve from Time Zero to Infinity (AUC [0-infinity]) of JNJ-64417184 | Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 72, 96, 120 hours postdose
  AUC (0-infinity) is the area under the plasma analyte concentration-time curve (AUC) from time zero to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z); wherein AUC (0-last) is area under the plasma concentration-time curve from time zero to last measurable concentration, C(last) is the last observed measurable (non-BQL) plasma analyte concentration; extrapolations of more than 20% of the total AUC are reported as approximations, and lambda(z) is apparent terminal elimination rate constant.
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 28 Days
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product does not necessarily have a causal relationship with the treatment. Therefore, it can be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to that medicinal product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- PRA Health Sciences Onderzoekscentrum Groningen, locatie Martini, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency